CLINICAL TRIAL: NCT00226122
Title: The Effect of Indomethacin in Monosymptomatic Enuresis Nocturnal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Konstantinos Kamperis MD PhD, Pediatric Research Laboratory, Aarhus University Hospital Skejby Aarhus Denmark
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: INDO181202; 01
Record Dates: First submitted 2005-09-23; First posted 2005-09-26 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Enuresis
Keywords: Enuresis; Nocturnal; Monosymptomatic; DDAVP; Indomethacin; Randomized
MeSH Terms: conditions — Enuresis | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Indomethacin — Indomethacin capsules 50 mg
  Other Names: Confortid

SUMMARY:
Monosymptomatic nocturnal enuresis, defined as the involuntary loss of urine during the night at an age where voluntary bladder control should have been attained and on the background of normal urinary tract function, is a rather common disease of childhood with an estimated prevalence of 5-10% at tha age of 7 and a spontaneous remission rate of 15% per year.

The present study consists of two phases; an in-patient phase and an ambulatory phase.

In the in-patient phase we will examine the regulation of sodium and the circadian rhythm of the hormones that affect this regulation in children with enuresis nocturnal and healthy children, as well as the impact of indomethacin on renal water and electrolyte excretion.

In the ambulatory phase we will examine the efficacy and safety of a treatment modality consisting of a combination of dDAVP and indomethacin in patients with severe enuresis where dDAVP as monotherapy is inadequate.

A significant number of children with enuresis and nocturnal polyuria do not respond to treatment with dDAVP. If a combination treatment with dDAVP and indomethacin proves superior to dDAVP alone the regimen could readily be used in those difficult to cure cases of enuresis.

DETAILED DESCRIPTION:
The "in-patient" phase is a comparative circadian study of three groups of participants and a non-placebo controlled study of the renal effects of indomethacin with special reference the renal handling of sodium.

The ambulatory phase is designed as a randomized double blind, crossover placebo controlled for indomethacin study of the efficacy and safety of a combination treatment with indomethacin and dDAVP.

In-patient phase: Primary effect parameters will be the diuresis, urinary osmolality, sodium excretion prior to and after the administration of indomethacin.

Secondary effect parameters will be the following: GFR, K+ excretion, creatinine excretion, urea excretion, as well as urinary concentrations of aquaporin 2 (AQP2), PGE2, AVP, URO, Na-transporter protein, concentration of renin, ANG II, ALDO, ANP, in plasma, prior to and after the administration of indomethacin.

Ambulatory phase: Primary effect parameter will be the number of dry nights achieved in the two treatment periods. Secondary effect parameters will be the nocturnal urine production, and the enuresis volumes In-patient phase: Day-night ratios will be calculated for all parameters tested. The circadian rhythm of hormones blood pressure and electrolyte excretion will be analyzed using COSINOR analysis.

The effect of indomethacin on the parameters tested will be compared to the basal measurements using student's t-test, ANOVA for repeated measurements or non-parametric tests. All statistical inference will take place on a "protocol population" basis.

Ambulatory phase: The efficacy of the combination treatment will be tested against placebo (only for indomethacin) with help of student's t-test, x2 test or non-parametric tests.

The results from the home recordings will be compared for the two treatment periods using non-parametric tests. The effect parameters that will undergo statistical analysis are the number of wet nights, the enuresis volume and the nocturnal urine production. The analysis will be on the basis of intention to treat population.

ELIGIBILITY:
Inclusion Criteria:

* Monosymptomatic enuresis nocturnal
* At least 3 nights with enuresis per week
* Incomplete response to dDAVP

Exclusion Criteria:

* Daytime incontinence
* Urgency
* Frequency
* Other conditions that influence normal urine production

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2003-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Enuresis episodes | 3 and 7 weeks

SECONDARY OUTCOMES:
Urine production, electrolyte excretion, hormonal changes | 3 and 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Kamperis, MD. PhD, Principal Investigator — Clinical Institute, University of Aarhus
Locations (1):
- Dept of Pediatrics, Aarhus University Hospital, Aarhus N, Jutland, Denmark

REFERENCES:
- [Derived] Hahn D, Stewart F, Raman G. Desmopressin for nocturnal enuresis in children. Cochrane Database Syst Rev. 2025 Jul 29;7(7):CD002112. doi: 10.1002/14651858.CD002112.pub2. PMID 40728007
- [Derived] Kamperis K, Hagstroem S, Faerch M, Mahler B, Rittig S, Djurhuus JC. Combination treatment of nocturnal enuresis with desmopressin and indomethacin. Pediatr Nephrol. 2017 Apr;32(4):627-633. doi: 10.1007/s00467-016-3536-9. Epub 2016 Oct 27. PMID 27787700